CLINICAL TRIAL: NCT03871972
Title: Safety and Efficacy of Umbilical Cord Blood Transfusion in Patients With Hutchinson-Gilford Progeria Syndrome
Brief Title: Umbilical Cord Blood Transfusion in Progeria Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Head of Rehabilitation Medicine Department, Professor, Principal Investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-12-031
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hutchinson-Gilford Progeria Syndrome
MeSH Terms: conditions — Progeria | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCB injection group (Experimental): This pilot study includes only 2 subjects who are enrolled by invitation. Both subjects are included in this single arm.
  Interventions: Drug: Umbilical Cord Blood Unit

INTERVENTIONS:
Drug: Umbilical Cord Blood Unit — 3 infusions of umbilical cord blood (UCB) unit (TNC > 2.0ⅹ107cells/kg) each 4 months apart and take oral Sirolimus (1 mg/m2/day) for 7 days (from 3 days before UCB infusion until 3 days after UCB infusion)
  Other Names: Oral Sirolimus

SUMMARY:
This is a pilot study on safety and efficacy of umbilical cord blood therapy for patients with Hutchinson Gilford Progeria syndrome (HGPS). This is an 1 year trial with 3 IV infusions (4 months apart from each infusion) of umbilical cord blood units with oral Sirolimus to see the safety and efficacy.

DETAILED DESCRIPTION:
This is a pilot study on safety and efficacy of umbilical cord blood therapy for patients with Hutchinson Gilford Progeria syndrome (HGPS). HGPS is a rare genetic disease where affected LMNA gene coding lamin A protein leads to premature aging and early death.

Teenagers with HGPS are in high risk of atherosclerosis and ischemic stroke, and these are major reason of mortality in HGPS.Currently, there are no definite cure for this rare genetic disease. Among the potential drugs under investigation, Lornafarnib (farnesyltransferase inhibitor) lowered the carotid-femoral pulse wave velocity (cfPWV) and also lowered mortality.

Stem cell therapy has proven its efficacy in progeria mouse model. We are trying to study safety and efficacy of umbilical cord blood therapy in human HGPS patients.

ELIGIBILITY:
This is a pilot study including 2 patients with HGPS.

Inclusion Criteria:

* those who were clinically and genetically diagnosed as Hutchinson-Gilford progeria syndrome

Exclusion Criteria:

* those who show definite hemorrhage or ischemia on brain MRI
* those who are affected with systemic infection during study enrolling period
* those who are not able to able to make consents to the study; those who are not accompanying any guardians
* those who were enrolled in other clinical trials within last 30 days
* those who are not appropriate according to laboratory criteria

  1. whose ALT/AST > 2 fold of normal limit
  2. whose serum creatinine > 1.5 fold of normal limit
  3. whose total bilirubin > 2 fold of normal limit
  4. whose total WBC count < 3000/mm3
  5. whose platelet count < normal lower limit
* those who are diagnosed with other malignancies
* those who are affected by other serious medical (cardiopulmonary, gastrointestinal, endocrinologic, etc.) conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Carotid-femoral pulse wave velocity at 48 weeks | 48 weeks after UCB infusion
  measured by carotid doppler ultrasonography
Change from baseline serum HDL cholesterol at 48 weeks | 48 weeks after UCB infusion
  taken on routine lab
Change from baseline weight at 48 weeks | 48 weeks after UCB infusion
  measured by bioimpedance analysis

SECONDARY OUTCOMES:
Ankle-brachial index | baseline, 48 weeks after UCB infusion
  measured by automatic blood pressure gauge
Body fat proportion | baseline, 48 weeks after UCB infusion
  taken by bioimpedance analysis
Range of motion | baseline, 48 weeks after UCB infusion
  measured manually
height | baseline, 48 weeks after UCB infusion
  measured by bioimpedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Min Young Kim, MD, PhD, Principal Investigator — CHA University
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No